CLINICAL TRIAL: NCT04429256
Title: Prosthetic Valve and Graft Endocarditis With Mycobacterium Chimaera: Diagnosis, Course of Disease, and Therapy Recommendations
Brief Title: Prosthetic Valve and Graft Endocarditis With Mycobacterium Chimaera
Status: Completed | Type: Observational
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Other Study IDs: Req-2020-00373;ch20Reuthebuch2
Record Dates: First submitted 2020-06-09; First posted 2020-06-12 (Actual); Last update posted 2023-11-21 (Actual); Status verified 2023-11

CONDITIONS: Mycobacterium Chimaera Infections
Keywords: cardiac bypass heater-cooler devices; cardiac surgery
MeSH Terms: interventions — Data Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: data collection — retrospective analysis of perioperative data collected from patient medical charts and from a telephone enquiry

SUMMARY:
Mycobacterium chimaera infections have occurred in post-cardiac surgery patients in association with contaminated cardiac bypass heater-cooler devices.

So far optimal therapeutical concepts are not clear. At the University Hospital Basel Mycobacterium chimaera- infected protheses are replaced to decrease pathogenic burden and to support antibiotic long- term treatment. This study is to analyze the efficacy of this therapeutic approach.

ELIGIBILITY:
Inclusion Criteria:

* Patients with Mycobacterium chimaera infections after cardiac surgery at University Hospital Basel

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with Mycobacterium chimaera infections after cardiac surgery at University Hospital Basel
Sampling Method: Non-Probability Sample
Enrollment: 7 (Actual)
Dates: Start 2020-04-10 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
summary of disease course in patients with Mycobacterium chimaera- infections after cardiac surgery | at baseline
  Descriptive statistical analysis of disease course in patients with Mycobacterium chimaera- infections after cardiac surgery
summary of therapeutic interventions in patients with Mycobacterium chimaera- infections after cardiac surgery | at baseline
  Descriptive statistical analysis of therapeutic interventions in patients with Mycobacterium chimaera- infections after cardiac surgery

CONTACTS AND LOCATIONS:
Overall Officials: Oliver Reuthebuch, Prof. Dr. med., Principal Investigator — Cardiac Surgery Clinic University Hospital Basel
Locations (1):
- Cardiac Surgery Clinic University Hospital Basel, Basel, Switzerland